CLINICAL TRIAL: NCT04341207
Title: COVID 19 - Epidemiology of SARS-CoV-2 and Mortality to Covid19 Disease Upon Hydroxychloroquine and Azithromycin Therapy in French Cancer Patients
Brief Title: Epidemiology of SARS-CoV-2 and Mortality to Covid19 Disease in French Cancer Patients
Acronym: ONCOVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001250-21; 2020/3078 (Other: CSET number)
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Cancer & COVID 19
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Advanced Cancer Patients with SARS-CoV-2 positive test & Covid19 symptoms
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin
- Cohort 2 (No Intervention): Advanced Cancer Patients with SARS-CoV-2 negative test & Covid19 symptoms. Patients with a chest CT-scan compatible with Covid19 disease shall be treated in part B.
- Cohort 3 (No Intervention): Advanced Cancer Patients with SARS-CoV-2 positive or negative test & no Covid19 symptoms
- Cohort 4 (Experimental): Advanced Cancer Patients with SARS-CoV-2 positive test AND chest CT-scan compatible with Covid19 disease & no Covid19 symptoms & Pretreated or with frail conditions following the HCSP definition
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 200 mg 3 times a day for 10 days
  Arms: Cohort 1; Cohort 4
Drug: Azithromycin — Azithromycin 500 mg on day 1 followed by 250 mg/day for 4 days
  Arms: Cohort 1

SUMMARY:
To determine the prevalence and the 3-months incidence of SARS-CoV-2 in cancer patients (Part A).

To evaluate the Covid-19 disease-specific mortality rate in cancer patients treated by hydroxychloroquine and azithromycin (Part B).

ELIGIBILITY:
Inclusion Criteria:

* All types of locally advanced and metastatic malignancy
* Male/female participants
* Age>18 y.o.
* Signed informed consent for participation in the study
* No restriction on Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) Performance Status
* Subject should not have received a prior systemic anti-viral treatment for Covid19 disease.

Exclusion Criteria:

* Patients with known hypersensitivity to hydroxychloroquine or chloroquine, azithromycin, erythromycin, or any other macrolide, ketolide or any of the excipients of the hydroxychloroquine and/or azithromycin-based specialty used.
* Severe hepatic impairment and patients with severe cholestasis.
* Patients with renal insufficiency with creatinine clearance < 40 mL/min.
* Combinations of drugs contraindicated in accordance with the approvals of the specialties used.
* Patients currently treated with Tamoxifen
* Patients already treated by hydroxychloroquine or azithromycin for Covid19 disease or currently treated with other antiviral drugs against coronavirus.
* Patients with known contra-indication to treatment with the study drug, including retinopathy, G6PD deficiency, QT prolongation and severe hepato-cellular insufficiency.
* Patients post allogeneic hematopoietic stem cell transplantation are eligible to the Part B treatments but the potential toxic effects of hydroxychloroquin and azithromycin on hematopoietic stem cells should be taken into consideration by prescribers.
* Pregnant or breastfeeding women. Women of childbearing potential (WOCBP, as defined in appendix 2) should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence and the 3-months incidence of SARS-CoV-2 in cancer patients | Up to 3 months
Covid-19 disease-specific mortality rate in cancer patients treated by hydroxychloroquine and azithromycin | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided